CLINICAL TRIAL: NCT05415462
Title: A Phase 3, Randomized, Stratified, Observer-blind, Active-Controlled Study to Evaluate the Immunogenicity and Safety of mRNA-1010 Seasonal Influenza Vaccine in Adults 18 Years and Older
Brief Title: A Study of mRNA-1010 Seasonal Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1010-P301
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Seasonal Influenza
MeSH Terms: interventions — mRNA-1010 influenza vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1010 (Experimental): Participants will receive a single dose of mRNA-1010 by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1010
- Fluarix Tetra (Active Comparator): Participants will receive a single dose of Fluarix Tetra by IM injection on Day 1.
  Interventions: Biological: Fluarix Tetra

INTERVENTIONS:
Biological: mRNA-1010 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1010
Biological: Fluarix Tetra — Sterile suspension for injection
  Other Names: Licensed quadrivalent inactivated seasonal influenza vaccine; Fluarix Quadrivalent
  Arms: Fluarix Tetra

SUMMARY:
The primary objectives of this study are to evaluate the humoral immunogenicity of mRNA-1010 relative to that of an active comparator against vaccine-matched influenza A and B strains at Day 29, and to evaluate the safety and reactogenicity of mRNA-1010.

ELIGIBILITY:
Inclusion Criteria:

* Investigator has assessed that the participant understands and is willing and physically able to comply with protocol mandated follow-up, including all procedures.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, and agreement to continue adequate contraception through 90 days following vaccine administration.

Exclusion Criteria:

* Participant has had close contact to someone with SARS-CoV-2 infection or COVID-19 as defined by the United States (US) CDC or has had a positive SARS-CoV-2 test in the past 10 days prior to the Screening Visit.
* Participant is acutely ill or febrile (temperature ≥38.0℃ [100.4°F]) 72 hours prior to or at the Screening Visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day screening window and will retain their initially assigned participant number.
* Participant has a history of a diagnosis or condition that, in the judgment of the investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA or influenza vaccines or any components of the mRNA or influenza vaccines, including egg protein.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 180 days prior to the Screening Visit (for corticosteroids, ≥10 milligrams (mg)/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study. Inhaled, nasal, and topical steroids are allowed.
* Participant has received any vaccine authorized or approved by local health agency ≤28 days prior to study injection (Day 1) or plans to receive a vaccine authorized or approved by local health agency within 28 days before or after the study injection.
* Participant is not aware whether they have received an influenza vaccine in the past 12 months or has received a seasonal influenza vaccine or any other investigational influenza vaccine within 180 days prior to Day 1.
* Participant has tested positive for influenza by local health authority-approved testing methods within 180 days prior to the Screening Visit.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6102 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- Argentina (11):
  - CEI -Centro de Estudios Infectológicos, Buenos Aires
  - Consultorios Médicos Dr. Doreski, Buenos Aires
  - Expertia S.A- Mautalen Salud e Investigacion, Buenos Aires
  - Fundación Socolinsky Centro de Vacunación Proteger, Buenos Aires
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Ciudad Autonoma Buenos Aires
  - Swiss Medical Center Barrio Parque, Ciudad Autónoma Buenos Aires
  - Sanatorio Allende S.A., Córdoba
  - Instituto Medico Platense, La Plata
  - Instituto Médico Río Cuarto, Río Cuarto
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
  - AES - AS - Clinica Mayo de Urgencias Medicas Cruz Blanca S.R.L. ("CLINICA MAYO") Tucumán, San Miguel de Tucumán
- Australia (14):
  - PARC Clinical Research, Adelaide
  - Paratus Clinical Research - Brisbane Clinic, Albion
  - Paratus Clinical Research - Western Sydney, Blacktown
  - Northern Beaches Clinical Research, Brookvale
  - Paratus Clinical Research - Canberra, Bruce
  - Emeritus Research, Camberwell
  - Monash Health, Monash Medical Centre, Clayton
  - Paratus Clinical Research - Central Coast, Kanwal
  - Australian Clinical Research Network, Maroubra
  - University of Melbourne, Parkville
  - University of the Sunshine Coast, Sippy Downs
  - Griffith University, Southport
  - AusTrials (Wellers Hill), Tarragindi
  - CMAX - Woodville, Woodville
- Colombia (16):
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Acacías, Acacías
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Aguazul, Aguazul
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Armenia, Armenia
  - Clinica de la Costa Ltda - PPDS, Barranquilla
  - Caja de Compensacion Familiar CAFAM sede Centro de atención en salud CAFAM Floresta, Bogotá
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Bogota, Bogotá
  - Unidad Integral de Endocrinologia, Bogotá
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Chia, Chía
  - Fundacion Oftalmologica de Santander Foscal, Floridablanca
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Girardot, Girardot
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Ibague, Ibagué
  - AES - AS - Centro de Investigación Clínica CIC S.A.S (CECIC) Medelin, Medellín
  - Clínica Universitaria Bolivariana, Medellín
  - Centro de Estudios en Infectología Pediatrica S.A.S - PPDS, Santiago de Cali
  - Fundación Hospital Universidad del Norte, Soledad
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Yopal, Yopal
- Panama (3):
  - Centro De Vacunacion Internacional, S.A. (Cevaxin) Sede La Chorrera, Panama City
  - CEVAXIN 24 de diciembre, Panama City
  - CEVAXIN Avenida México, Panama City
- Philippines (9):
  - Asian Hospital and Medical Center, City of Muntinlupa
  - Healthlink Iloil, Iloilo City
  - St. Paul's Hospital, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Health Cube Medical Clinics, Mandaluyong
  - Manila Doctors Hospital, Manila
  - Medical Center Manila, Manila
  - San Juan de Dios Hospital, Pasay
  - Lung Center of The Philippines, Quezon City

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluarix Tetra: Participants received a single dose of Fluarix Tetra by intramuscular (IM) injection on Day 1.
- mRNA-1010: Participants received a single dose of mRNA-1010 by IM injection on Day 1.
Period: Overall Study
Arm/Group | Fluarix Tetra | mRNA-1010
Started | 3057 | 3045
Received Injection | 3048 | 3035
Completed | 2824 | 2857
Not Completed | 233 | 188
Not completed — Death | 18 | 10
Not completed — Lost to Follow-up | 72 | 64
Not completed — Physician Decision | 5 | 5
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Subject | 129 | 101
Not completed — Other Than Specified | 8 | 8

BASELINE CHARACTERISTICS:
Population: The Randomization Set included all participants who were randomly assigned to treatment, regardless of the participants' vaccination status in the study.
Groups:
- Fluarix Tetra: Participants received a single dose of Fluarix Tetra by IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Fluarix Tetra | mRNA-1010 | Total
Number analyzed (Participants) | 3057 | 3045 | 6102
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (16.49) | 48.0 (16.41) | 48.0 (16.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1742 | 1787 | 3529
  Male | 1315 | 1258 | 2573
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2222 | 2209 | 4431
  Not Hispanic or Latino | 812 | 819 | 1631
  Unknown or Not Reported | 23 | 17 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 1745 | 1733 | 3478
  Race: Black or African American | 18 | 15 | 33
  Race: Asian | 706 | 708 | 1414
  Race: American Indian or Alaska Native | 320 | 305 | 625
  Race: Native Hawaiian or Other Pacific Islander | 3 | 10 | 13
  Race: Multiple | 216 | 220 | 436
  Race: Other | 2 | 3 | 5
  Race: Not Reported | 3 | 3 | 6
  Race: Unknown | 42 | 46 | 88
  Race: Missing | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies at Day 29, as Measured by Hemagglutination Inhibition (HAI) Assay for Vaccine-matched Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
Time Frame: Day 29
Population: The Per Protocol Immunogenicity Set (PPIS) included all randomized participants who received any study vaccination, who had baseline and Day 29 antibody assessment via HAI assay, complied with the immunogenicity testing schedule, and had no significant protocol deviations that impacted key or critical data. Number Analyzed = participants evaluable for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 2823 | 2850
titer
  Influenza A H1N1 Antibody: number analyzed (Participants) | 2801 | 2831
  Influenza A H1N1 Antibody | 266.52 [256.16 to 277.29] | 268.94 [259.28 to 278.95]
  Influenza A H3N2 Antibody | 175.06 [167.61 to 182.85] | 290.19 [277.90 to 303.02]
  Influenza B/ Victoria Lineage: number analyzed (Participants) | 2801 | 2831
  Influenza B/ Victoria Lineage | 127.50 [122.13 to 133.11] | 84.16 [80.66 to 87.80]
  Influenza B/ Yamagata Lineage: number analyzed (Participants) | 2821 | 2850
  Influenza B/ Yamagata Lineage | 254.38 [245.52 to 263.57] | 169.98 [164.41 to 175.74]
Statistical Analysis 1: Comparison: Fluarix Tetra vs mRNA-1010; GMR (mRNA-1010 vs Fluarix) for Influenza A H1N1 Antibody; Test type: Non-Inferiority — The endpoint was tested for noninferiority of mRNA-1010 vs Fluarix for Influenza A H1N1 strain at a 2-sided 0.025 level; Geometric Mean Ratio (GMR) = 1.010, 97.5% CI 2-sided [0.952 to 1.071]
Statistical Analysis 2: Comparison: Fluarix Tetra vs mRNA-1010; GMR (mRNA-1010 vs Fluarix) for Influenza A H3N2 Antibody; Test type: Non-Inferiority — The endpoint was tested for noninferiority of mRNA-1010 vs Fluarix for Influenza A H3N2 strain at a 2-sided 0.025 level; GMR = 1.657, 97.5% CI 2-sided [1.562 to 1.757]
Statistical Analysis 3: Comparison: Fluarix Tetra vs mRNA-1010; GMR (mRNA-1010 vs Fluarix) for Influenza B/ Victoria Lineage; Test type: Non-Inferiority — The endpoint was tested for noninferiority of mRNA-1010 vs Fluarix for Influenza B Victoria-lineage strain at a 2-sided 0.025 level; GMR = 0.665, 97.5% CI 2-sided [0.630 to 0.702]
Statistical Analysis 4: Comparison: Fluarix Tetra vs mRNA-1010; GMR (mRNA-1010 vs Fluarix) for Influenza B/ Yamagata Lineage; Test type: Non-Inferiority — The endpoint was tested for noninferiority of mRNA-1010 vs Fluarix for Influenza B Yamagata-lineage strain at a 2-sided 0.025 level; GMR = 0.661, 97.5% CI 2-sided [0.630 to 0.693]

2. Primary Outcome: Percentage of Participants Reaching Seroconversion at Day 29, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
  Seroconversion was defined as either a Baseline HAI titer <1:10 and a post-Baseline titer ≥1:40 or a Baseline HAI titer ≥1:10 and a minimum 4-fold rise in post-Baseline HAI Ab titer.
Time Frame: Day 29
Population: The PPIS included all randomized participants who received any study vaccination, who had baseline and Day 29 antibody assessment via HAI assay, complied with the immunogenicity testing schedule, and had no significant protocol deviations that impacted key or critical data. Number Analyzed = participants evaluable for specified categories.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 2823 | 2850
percentage of participants
  Influenza A H1N1 Antibody: number analyzed (Participants) | 2801 | 2831
  Influenza A H1N1 Antibody | 70.6 [68.89 to 72.30] | 76.4 [74.76 to 77.92]
  Influenza A H3N2 Antibody | 63.2 [61.35 to 64.94] | 80.1 [78.56 to 81.52]
  Influenza B/ Victoria Lineage: number analyzed (Participants) | 2801 | 2831
  Influenza B/ Victoria Lineage | 49.7 [47.83 to 51.57] | 32.4 [30.63 to 34.11]
  Influenza B/ Yamagata Lineage: number analyzed (Participants) | 2821 | 2850
  Influenza B/ Yamagata Lineage | 65.2 [63.36 to 66.91] | 49.5 [47.62 to 51.33]
Statistical Analysis 1: Comparison: Fluarix Tetra vs mRNA-1010; Percentage Difference (mRNA-1010 vs Fluarix) for Influenza A H1N1 Antibody; Test type: Non-Inferiority — The endpoint was tested for noninferiority of mRNA-1010 vs Fluarix for Influenza A H1N1 strain at a 2-sided 0.025 level; Percentage Difference = 5.75, 97.5% CI 2-sided [3.12 to 8.38]
Statistical Analysis 2: Comparison: Fluarix Tetra vs mRNA-1010; Percentage Difference (mRNA-1010 vs Fluarix) for Influenza A H3N2 Antibody; Test type: Non-Inferiority — The endpoint was tested for noninferiority of mRNA-1010 vs Fluarix for Influenza A H3N2 strain at a 2-sided 0.025 level; Percentage Difference = 16.91, 97.5% CI 2-sided [14.27 to 19.54]
Statistical Analysis 3: Comparison: Fluarix Tetra vs mRNA-1010; Percentage Difference (mRNA-1010 vs Fluarix) for Influenza B/Victoria Lineage; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 3]; Percentage Difference = -17.34, 97.5% CI 2-sided [-20.22 to -14.43]
Statistical Analysis 4: Comparison: Fluarix Tetra vs mRNA-1010; Percentage Difference (mRNA-1010 vs Fluarix) for Influenza B/Yamagata Lineage; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 4]; Percentage Difference = -15.68, 97.5% CI 2-sided [-18.57 to -12.76]

3. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were collected in an electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. All solicited ARs considered causally related to injection were graded 0-4 (per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials); lower score indicates lower severity, and a higher score indicates greater severity. Note, not all solicited ARs were considered adverse events (AEs). The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: 7 days post-vaccination
Population: The Solicited Safety Set included all randomized participants who received any study vaccination and contributed any solicited AR data, that is, had at least 1 post-baseline solicited safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 3046 | 3035
Participants
  Any | 1463 | 2137
  Grade 1 | 1051 | 1160
  Grade 2 | 309 | 659
  Grade 3 | 93 | 312
  Grade 4 | 10 | 6

4. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. Number of participants with unsolicited AEs (SAEs and non-serious AEs) up to 28 days post-vaccination are reported in this outcome measure.
Time Frame: Up to 28 days post-vaccination
Population: The Safety Set included all participants who were randomized and received any study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 3048 | 3035
Participants | 749 | 800

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Discontinuation
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that lead to an unscheduled visit to an healthcare practitioner. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or coronavirus disease 2019 [COVID-19] and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). Number of participants with SAEs, AESIs, MAAEs, and AEs leading to discontinuation up to the end of study (Day 361) are reported in this outcome measure.
Time Frame: Day 1 through Day 361 (Month 12)
Population: The Safety Set included all participants who were randomized and received any study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 3048 | 3035
Participants
  SAEs | 131 | 132
  AESIs | 13 | 9
  MAAEs | 1481 | 1422
  AEs Leading to Discontinuation | 17 | 10

6. Secondary Outcome: Number of Participants With First Episode of Reverse Transcription Polymerase Chain Reaction (RT-PCR)-Confirmed Protocol-Defined Influenza-Like Illness (ILI) Caused by Any Strain of Influenza Virus
Description: A protocol-defined ILI was determined by the occurrence of at least 1 respiratory illness symptom concurrently with at least 1 systemic symptom, or the occurrence of any 2 or more respiratory symptoms. Respiratory symptoms included sore throat, cough/rhinorrhea/nasal congestion (≥1 of the 3 symptoms count as 1 respiratory symptom), sputum production, wheezing, or difficulty breathing. Systemic symptoms included body temperature >37.2 degrees Celsius (°C) (>99 degrees Fahrenheit [°F]), chills, tiredness, headache, myalgia, nausea/vomiting, or diarrhea.
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: The Modified Intent-to-Treat (mITT) Set included all participants who were randomized and received any study vaccination and who provided any follow-up for ILI beginning at least 14 days following administration of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 2979 | 2980
Participants | 54 | 64

7. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed Centers for Disease Control and Prevention (CDC)-Defined ILI Caused by Any Strain of Influenza Virus
Description: A CDC-defined ILI was defined as body temperature ≥37.8°C (100°F) accompanied by cough and/or sore throat.
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: The mITT Set included all participants who were randomized and received any study vaccination and who provided any follow-up for ILI beginning at least 14 days following administration of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 2979 | 2980
Participants | 22 | 24

8. Secondary Outcome: Number of Participants With First Episode of RT-PCR-Confirmed Protocol-Defined ILI Caused by Any Strain of Influenza Virus in Participants Aged 50 Years and Older or 65 Years and Older
Description: A protocol-defined ILI was determined by the occurrence of at least 1 respiratory illness symptom concurrently with at least 1 systemic symptom, or the occurrence of any 2 or more respiratory symptoms. Respiratory symptoms included sore throat, cough/rhinorrhea/nasal congestion (≥1 of the 3 symptoms count as 1 respiratory symptom), sputum production, wheezing, or difficulty breathing. Systemic symptoms included body temperature >37.2°C (>99°F), chills, tiredness, headache, myalgia, nausea/vomiting, or diarrhea.
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: The mITT Set included all participants who were randomized and received any study vaccination and who provided any follow-up for ILI beginning at least 14 days following administration of study intervention. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 1534 | 1512
Participants
  50 Years and Older | 15 | 21
  65 Years and Older: number analyzed (Participants) | 580 | 573
  65 Years and Older | 3 | 5

9. Secondary Outcome: Percentage of Participants With HAI Titer ≥ 1:40 at Day 29
Description: as for outcome 1
Time Frame: Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 2823 | 2850
percentage of participants
  Influenza A H1N1 Antibody: number analyzed (Participants) | 2801 | 2831
  Influenza A H1N1 Antibody | 97.0 [96.30 to 97.60] | 97.6 [97.00 to 98.16]
  Influenza A H3N2 Antibody | 92.1 [91.04 to 93.07] | 96.9 [96.21 to 97.52]
  Influenza B/Victoria Lineage: number analyzed (Participants) | 2801 | 2831
  Influenza B/Victoria Lineage | 88.0 [86.78 to 89.22] | 80.7 [79.25 to 82.19]
  Influenza B/Yamagata Lineage: number analyzed (Participants) | 2821 | 2850
  Influenza B/Yamagata Lineage | 98.5 [97.99 to 98.92] | 96.7 [95.94 to 97.29]

10. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-HA Antibodies at Day 29, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% confidence interval (CI) for GMFR was calculated based on the t distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Baseline, Day 29
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluarix Tetra | mRNA-1010
Number analyzed (Participants) | 2823 | 2850
ratio
  Influenza A H1N1 Antibody: number analyzed (Participants) | 2801 | 2831
  Influenza A H1N1 Antibody | 7.27 [6.93 to 7.62] | 7.42 [7.13 to 7.73]
  Influenza A H3N2 Antibody | 4.92 [4.73 to 5.12] | 8.15 [7.83 to 8.48]
  Influenza B/Victoria Lineage: number analyzed (Participants) | 2801 | 2831
  Influenza B/Victoria Lineage | 3.59 [3.44 to 3.73] | 2.38 [2.30 to 2.46]
  Influenza B/Yamagata Lineage: number analyzed (Participants) | 2821 | 2850
  Influenza B/Yamagata Lineage | 5.27 [5.07 to 5.48] | 3.46 [3.35 to 3.56]

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were collected throughout the entire period of the study (from Day 1 up to the end of study [Day 361]). Other (not including serious) adverse events were collected for 28 days after the vaccination.
Description: As pre-specified, All-cause mortality data were collected and reported for all randomized participants; and Serious and Non-serious adverse events data were collected and reported for all randomized participants who received the study drug. Adverse event data were collected during the study visit by the investigator. A participant may experience the same event both as SAE and non-SAE.
Groups:
- Fluarix Quadrivalent 60 ug: Participants received a single intramuscular (IM) injection of Fluarix Quadrivalent 60 ug on Day 1
- mRNA-1010 50 ug: Participants received a single intramuscular (IM) injection of mRNA-1010 50 ug on Day 1
Arm/Group | Fluarix Quadrivalent 60 ug | mRNA-1010 50 ug
All-Cause Mortality (participants affected / at risk) | 18/3057 | 10/3045
Serious Adverse Events (participants affected / at risk) | 131/3048 | 132/3035
Other Adverse Events (participants affected / at risk) | 809/3048 | 803/3035
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Quadrivalent 60 ug (N=3048) | mRNA-1010 50 ug (N=3035)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Amoebic colitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacillus bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 3 (3) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Leptospirosis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 9 (9)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 4 (4)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Spleen tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 12 (12)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 2 (2)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (4) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 4 (4)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial injury (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spigelian hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 7 (7) | 7 (7)
Cholestasis of pregnancy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Dehiscence (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Quadrivalent 60 ug (N=3048) | mRNA-1010 50 ug (N=3035)
COVID-19 (Infections and infestations) | 424 (445) | 442 (461)
Rhinovirus infection (Infections and infestations) | 150 (167) | 167 (185)
Upper respiratory tract infection (Infections and infestations) | 205 (243) | 200 (251)
Influenza like illness (General disorders) | 168 (207) | 165 (206)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT05415462/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT05415462/SAP_001.pdf